CLINICAL TRIAL: NCT05127980
Title: Occurrence of Antibodies Cross-reacting With Autoantigens in Primary EBV Infection - a Longitudinal, Observational Study
Brief Title: Occurrence of Antibodies Cross-reacting With Autoantigens in Primary EBV Infection
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-01338; am21Osthoff2
Record Dates: First submitted 2021-10-25; First posted 2021-11-19 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Epstein-Barr Virus (EBV) Infection
Keywords: Infectious mononucleosis (IM); Viral capsid antigen (VCA); EBV nucleic antigen (EBNA); Systemic lupus erythematosus (SLE); Chronic fatigue syndrome (CFS); cross-reacting antibodies; molecular mimicry
MeSH Terms: conditions — Epstein-Barr Virus Infections; Infections; Infectious Mononucleosis; Lupus Erythematosus, Systemic; Fatigue Syndrome, Chronic | interventions — Procalcitonin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and serum samples will be coded by a study nurse and stored at -80°C in a dedicated freezer with limited access to unauthorized personal for future research projects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with confirmed primary EBV infection: 40 patients with confirmed primary EBV infection as confirmed by the treating clinician and defined by:
  - Compatible clinical (infectious mononucleosis symptoms including but not limited to malaise, headache, fever, tonsillitis, pharyngitis, cervical lymph nodes enlargement) and laboratory picture (lymphocyte count elevation, LUC cells, reactive lymphocytes in manual differential, elevated liver enzymes; of note, not all typically described features have to be fulfilled)
  AND
  - serology compatible with primary EBV infection (anti-EBNA IgG negative, anti-VCA IgG negative, anti-VCA IgM positive OR anti-EBNA IgG negative, anti-VCA IgG positive, anti- VCA IgM positive)
  Interventions: Other: Data collection: Participant characteristics (Illness course, complications of primary EBV infection and provided treatments); Other: Data collection: blood samples (analysed for EBV serology, auto-antibody-testing/biobanking, RNA expression analyses, procalcitonin); Other: Data collection: Patient reported outcome (Fatigue questionnaires)
- control patients: 40 control patients (Clinical picture of upper respiratory tract infection (including but not limited to tonsillitis/pharyngitis, malaise, headache, cough, rhinitis, cervical node enlargement)) and/ or confirmed primary Cytomegalovirus (CMV) infection
  Interventions: Other: Data collection: Participant characteristics (Illness course, complications of primary EBV infection and provided treatments); Other: Data collection: blood samples (analysed for EBV serology, auto-antibody-testing/biobanking, RNA expression analyses, procalcitonin); Other: Data collection: Patient reported outcome (Fatigue questionnaires)

INTERVENTIONS:
Other: Data collection: Participant characteristics (Illness course, complications of primary EBV infection and provided treatments) — Data collection: Participant characteristics (Illness course, complications of primary EBV infection and provided treatments) during 12 months (baseline visit and follow-up visits at 3, 6 and 12 months).
Other: Data collection: blood samples (analysed for EBV serology, auto-antibody-testing/biobanking, RNA expression analyses, procalcitonin) — Data collection: blood samples (analysed for EBV serology, auto-antibody-testing/biobanking, RNA expression analyses, procalcitonin) during 12 months (baseline visit and follow-up visits at 3, 6 and 12 months).
Other: Data collection: Patient reported outcome (Fatigue questionnaires) — Data collection: Patient reported outcome (Fatigue questionnaires) at 6 and 12 months.

SUMMARY:
The aim of this study is to assess the occurrence of antibodies cross-reacting with autoantigens that have been detected in the context of SLE in patients with primary EBV infection over time compared to a control group. It is to establish a biobank of patients with primary EBV infection allowing to longitudinally analyze the immune response and its accompanying inflammatory processes with focus on the occurrence of antibodies cross-reacting with autoantigens associated with SLE and other autoimmune diseases.

Substudies will analyze

* characteristics of primary EBV infection patients treated with antibiotics in comparison to patients treated without antibiotics and outcomes of these treatment regimens (occurrence of acute complications such as peritonsillar abscess (PTA) or need for tonsillectomy, frequency of fatigue or symptoms associated with chronic fatigue syndrome).
* Procalcitonin (PCT) concentrations in primary EBV infection compared to control patients with similar symptoms and its association with disease severity and local complications.
* the occurrence of fatigue and symptoms associated with chronic fatigue syndrome 6 and 12 months after primary EBV infection.

DETAILED DESCRIPTION:
Epstein-Barr Virus (EBV) is a lymphotropic herpes virus and the causative agent of infectious mononucleosis (IM). The course of EBV infection is determined by the virus load and an individuals' immune system state, which in turn is determined by the person's gene composition, other infection history and several environmental factors, which all may influence the immune capacity of a person to various degrees. Many diseases are known to be associated with EBV infection, among those diseases are systemic autoimmune diseases. With regard to EBV, prior infection with the virus seems to be of crucial importance for the development of systemic lupus erythematosus (SLE). Autoantibodies against complement C1q (anti-C1q) can be induced in vivo by the Epstein-Barr virus-derived antigenic site 'EBNA348' (also being part of the C-terminal EBNA-1).

This study is to analyze whether the primary infection with EBV (leading to IM and antibodies targeting EBV-derived antigens including antibodies against EBNA-1) leads to an at least transient occurrence of antibodies against the virus that have the potential to cross-react with autoantigens as described in patients with systemic autoimmune diseases (e.g. complement C1q, dsDNA, Ro, Sm, MOG, NF186 and others). The advantage of an analysis of patients with primary infection is that the de novo synthesis of antibodies against the virus will allow to determine the time-dependent evolution of the antibody repertoire against the virus as well as against a number of autoantigens.

ELIGIBILITY:
Inclusion Criteria:

Participants fulfilling all of the following inclusion criteria are eligible for the infectious mononucleosis (IM) group:

* Informed consent as documented by signature
* Confirmed primary EBV infection as confirmed by the treating clinician and defined by:
* Compatible clinical (infectious mononucleosis symptoms including but not limited to malaise, headache, fever, tonsillitis, pharyngitis, cervical lymph nodes enlargement) and laboratory picture (lymphocyte count elevation, LUC cells, reactive lymphocytes in manual differential, elevated liver enzymes; of note, not all typically described features have to be fulfilled)

AND

* serology compatible with primary EBV infection (anti-EBNA IgG negative, anti-VCA IgG negative, anti-VCA IgM positive OR anti-EBNA IgG negative, anti-VCA IgG positive, anti- VCA IgM positive).

Participants fulfilling all of the following inclusion criteria will be eligible for the control group:

* Informed consent as documented by signature.
* one of the following:

  1. Clinical picture of upper respiratory tract infection (including but not limited to tonsillitis/pharyngitis, malaise, headache, cough, rhinitis, cervical node enlargement)
  2. confirmed primary Cytomegalovirus (CMV) infection (an optimal control group; however, the number of patients with a diagnosis of primary CMV infection is limited).

Exclusion Criteria:

* Suspicion/diagnosis of IM as per judgement of the treating clinician (control group only); this individual may be eligible later for the IM group if primary EBV infection is confirmed, subsequently.
* Immunosuppression (broadly defined as primary/secondary immunodeficiency or treatment with an immunosuppressive medication including ≥ 10mg prednisone equivalent).
* History of autoimmune disease (e.g. SLE, vasculitis etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients and outpatients with symptoms of infectious mononucleosis (IM) or a sore throat who are treated at the University Hospital of Basel will be approached.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in occurrence of antibodies cross-reacting with autoantigens in patients with primary EBV infection | at Visit 2 (day 1 (+ 1 day)), Visit 3 (3 months +/- 21 days), Visit 4 (6 months +/- 1 month) and Visit 5 (12 months +/-2 months)
  Change in occurrence of antibodies cross-reacting with autoantigens in patients with primary EBV infection compared to a control group.

SECONDARY OUTCOMES:
Change in RNA expression profiles of peripheral blood cells | at Visit 2 (day 1 (+ 1 day)), Visit 3 (3 months +/- 21 days), Visit 4 (6 months +/- 1 month) and Visit 5 (12 months +/-2 months)
  Change in RNA expression profiles of peripheral blood cells in patients with primary EBV infection over time and compared to a control group.
Change in Fatigue Assessment Scale (FAS) | at month 6 and at month 12
  The total score ranges from 10 to 50. A total FAS score < 22 indicates no fatigue, a score ≥ 22 indicates fatigue.
Change in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) questionnaire | at month 6 and at month 12
  FACIT-F is a 13-item instrument designed to assess fatigue/ tiredness and its impact on daily activities and functioning in a number of chronic diseases. The instrument includes items such as tiredness, weakness, listlessness, lack of energy, and the impact of these feelings on daily functioning (e.g., sleeping, and social activities). Items are scored on a 0 - 4 response scale with anchors ranging from "Not at all" to "Very much so" (in which higher scores represent better functioning or less fatigue).
Change in Procalcitonin (PCT) (Substudy Procalcitonin) | on day 1 and day 3 (+/-1 day)
  Change in PCT compared in primary EBV infection patients with different disease severities and different treatment modalities (in particular if they received antibiotics or not), and in comparison to a control group (with mostly (viral) upper respiratory tract infection or primary CMV infection); In IM and control patients admitted to hospital, blood will be collected for PCT measurement
Occurrence of acute complications such as PTA or need for tonsillectomy | at Visit 2 (day 1 (+ 1 day)) and Visit 3 (3 months +/- 21 days),
  Occurrence of acute complications such as PTA or need for tonsillectomy in primary EBV infection patients treated with antibiotics in comparison to patients treated without antibiotics

CONTACTS AND LOCATIONS:
Overall Officials: Michael Osthoff, PD Dr. med., Principal Investigator — University Hospital Basel, Division of Internal Medicine
Locations (1):
- University Hospital Basel, Division of Internal Medicine, Basel, Switzerland